CLINICAL TRIAL: NCT07270367
Title: Finerenone and Cardiac Remodeling: A Randomized, Double- Blind, Placebo-Controlled Study to Evaluate The Effects of Finerenone on Ventricular Remodeling
Brief Title: Finerenone and Cardiac Remodeling
Acronym: FINE-MECH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Subodh Verma (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Subodh Verma, Professor of Surgery and Pharmacology & Toxicology, Canadian Medical and Surgical Knowledge Translation Research Group
Organization: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-0011
Record Dates: First submitted 2025-11-13; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Finerenone; Left Ventricle Remodeling; Double-blind; Randomized; Heart Failure; Multicentre; Cardiorenal
MeSH Terms: conditions — Heart Failure; Ventricular Remodeling | interventions — finerenone

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, randomized (1:1), placebo-controlled trial of finerenone vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Active Comparator): Active treatment group
  Interventions: Drug: Finerenone
- Placebo (Placebo Comparator): Control treatment group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finerenone — Participants will be allocated a starting dose of 10 or 20 mg of finerenone (dependent on kidney function) once daily, in addition to standard-of-care. Participants may be up-titrated or down-titrated based on potassium levels or estimated glomerular filtration rate with a minimum dose of 10 mg and maximum dose of 40 mg finerenone
  Other Names: Kerendia
  Arms: Finerenone
Drug: Placebo — Participants will be allocated a starting dose of 10 or 20 mg of placebo (dependent on kidney function) once daily, in addition to standard-of-care. Participants may be up-titrated or down-titrated based on potassium levels or estimated glomerular filtration rate with a minimum dose of 10 mg and maximum dose of 40 mg placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug finerenone (Karendia) can improve heart function in participants who are at risk for heart and kidney disease.

The main question it aims to answer is whether adding finerenone to standard-of-care heart failure medical therapies will beneficially alter the heart structure and function of people who have risk factors for heart and kidney complications and whose left side of the heart is enlarged.

The researchers will compare finerenone to a placebo (a look-alike substance that contains no drug) to see if finerenone improves heart structure and function.

Participants will:

* take a finerenone or a placebo tablet once a day for 12 months
* have a cardiac magnetic resonance imaging (cMRI; a safe, non-invasive scan to measure heart mass, stiffness and function) test at the beginning of the study and 12 months later
* visit the clinic after one, three, six and twelve months to assess overall health and/or perform blood or urine tests

DETAILED DESCRIPTION:
Finerenone is a potent and selective oral non-steroidal mineralocorticoid receptor antagonist that has demonstrated marked cardiovascular benefits in people living with diabetic kidney disease, heart failure with mildly reduced ejection fraction, and heart failure with preserved ejection fraction. However, the mechanistic basis of these broad cardiovascular benefits remains unclear.

The FINE-MECH CardioLink-11 trial is a multicentre, prospective, randomized, double-blind trial of finerenone vs placebo in addition to standard-of-care in adults with evidence of left ventricular hypertrophy and cardiorenal risk factors. A total of 156 individuals who provide written informed consent and meet all the inclusion criteria (and none of the exclusion criteria) will be assigned (1:1) to receive either finerenone or placebo QD for 12 months. There will be 6-7 clinic visits. Outcome assessors will be blinded to the investigational product allocation and the time point at which each assessment was completed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥18 years of age who are willing and able to provide signed informed consent
* Evidence of left ventricular (LV) hypertrophy ≤12 months prior to or at screening showing at least one (≥1) of the following:

  1. Interventricular septal (IVS) thickness by echocardiography: Female ≥1.2 cm or Male ≥1.3 cm
  2. Posterior wall (PW) thickness by echocardiography: Female ≥1.2 cm or Male ≥1.3 cm
  3. Left ventricular mass indexed to baseline body surface area (LVMi) by echocardiography: Female >95 g⁄m^2 or Male >115 g⁄m^2
  4. LVMi (with papillary muscles included in the LV blood pool) by cMRI: Female >59 g⁄m^2 or Male >75 g⁄m^2
  5. LVMi (if the papillary muscles are included in the LVM) by cMRI: Female >68 g⁄m^2 or Male >85 g⁄m^2
* The presence of at least one (≥1) of the following risk factors:

  1. History of heart failure with preserved ejection fraction (left ventricular ejection fraction [LVEF] ≥50%);
  2. Type 2 diabetes mellitus;
  3. Estimated glomerular filtration rate (eGFR) ≥25 and <75 mL/min/1.73 m^2;
  4. Urine albumin-creatinine ratio (UACR) >3.39 mg/mmol and <565 mg/mmol;
  5. Left atrial volume indexed to baseline body surface area (LAVi) >40 mL/m^2 (by echocardiography and as measured by either the biplane area-length method or Simpson's biplane method);
  6. IVS ≥1.4 cm;
  7. PW ≥1.4 cm;
  8. LVMi ≥125 g⁄m^2 for males and ≥105 g⁄m^2 for females (by echocardiography);
  9. N-terminal pro-B-type natriuretic peptide (NT-proBNP; within past 6 months) ≥150 pg/mL if in sinus rhythm or ≥450 pg/mL if atrial fibrillation is present.
  10. Females who are of childbearing age can only be included if I. they are postmenopausal (i.e. no menstruation for at least one [≥1] year) or have had a surgical procedure ≥6 months at screening that prevents them from becoming pregnant; or II. the result of their pregnancy test at the baseline visit is negative, and they agree to use medically acceptable contraception methods to avoid pregnancy for the duration of the trial and for 1 month after taking the last dose of the assigned investigational product.

Exclusion Criteria:

* Females who are planning to become pregnant, are breastfeeding or are planning to breastfeed;
* Males who are planning to either father a child or donate sperm for the duration of the trial and for 1 month after taking the last dose of the assigned IP;
* Serum potassium level ≥5 mmol/L at the time of screening;
* eGFR <25 mL/min/1.73 m^2 at the time of screening or on kidney replacement therapy;
* UACR ≥565 mg/mmol at the time of screening;
* Seated systolic blood pressure <110 mmHg at the time of screening;
* History of pulmonary arterial hypertension;
* Type 1 diabetes mellitus;
* Body mass index ≥40 kg/m^2;
* Contraindication or inability to undergo MRI;
* Known persistent hypoalbuminemia (≤30 g/L on >1 measurement within last 6 months);
* Currently on a mineralocorticoid receptor antagonist (MRA) or in the opinion of the investigator, an MRA is either clinically indicated or contraindicated (e.g. history of marked hyperkalemia, marked hemodynamic stress, intolerance to MRAs) - individuals who previously experienced gynecomastia with spironolactone may be eligible if they meet all the inclusion criteria and none of the exclusion criteria;
* Requirement of any intravenous (IV) vasodilating drug (e.g. nitrates, nitroprusside), any IV natriuretic peptide (e.g. nesiritide, carperitide), any IV positive inotropic agents, or mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device) ≤24 hours prior to randomization;
* Concomitant systemic therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors (e.g. itraconazole, ritonavir, indinavir, cobicistat, clarithromycin) or moderate or potent CYP3A4 inducers, that cannot be discontinued 7 days prior to randomization and for the duration of the treatment period;
* History of cardiac device implant (e.g. implantable cardioverter defibrillator/cardiac resynchronization therapy/pacemaker) or planned device implant ≤90 days after screening;
* Hospitalized for heart failure (HF) requiring initiation or change in HF therapy or an urgent visit for HF requiring IV diuretic therapy, either ≤45 days prior to screening;
* LVEF <40% per the most current echocardiogram or MRI;
* Symptomatic bradycardia or second- or third-degree heart block without a pacemaker;
* History of peripartum cardiomyopathy, chemotherapy-induced cardiomyopathy, viral myocarditis, right HF in the absence of left-sided structural disease, pericardial constriction, hypertrophic cardiomyopathy, or infiltrative cardiomyopathy including amyloidosis;
* Myocardial infarction ≤45 days of screening;
* Planned or previous cardiac surgery or major non-cardiac surgery ≤45 days of screening;
* Planned or previous percutaneous coronary intervention ≤45 days of screening;
* Stroke or transient ischemic stroke ≤90 days before randomization;
* Severe valvular heart disease;
* Addison's disease;
* Individuals who are heart or kidney transplant recipients or who are (or are expected to be) listed for heart transplant, kidney dialysis or a kidney transplant ≤12 months of screening;
* Any other known condition or therapy which would make the individual unsuitable for this trial (e.g. hepatic insufficiency, liver biomarkers >3X upper limit of normal, chronic pulmonary disease, life threatening arrhythmia, uncontrolled arrhythmia) or not allow participation for the full planned trial duration (e.g. active malignancy ≤24 months of screening or condition limiting life expectancy to <12 months);
* Allergy to finerenone (or its excipients);
* Allergy to gadolinium;
* Participation in an investigational study ≤15 days prior to screening, or during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass indexed to baseline body surface area (LVMi) | 12 months
  Change in LVMi (g/m^2), measured by cardiac magnetic resonance imaging (cMRI) from baseline to 12 months of treatment with finerenone compared to placebo. cMRI evaluations will be made from standard 2D views with and without gadolinium as a contrast agent. All acquired sequences will adhere to the current clinical standard of care.

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | 12 months
  Change in LVEF, measured by cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Left Ventricular End-Diastolic Volume indexed to baseline body surface area (LVEDVi) | 12 months
  Change in LVEDVi, measured by cMRI and indexed to baseline body surface area, from baseline to 12 months of treatment with finerenone compared to placebo.
Left Ventricular End-Systolic Volume indexed to baseline body surface area (LVESVi) | 12 months
  Change in LVESVi, measured by cMRI and indexed to baseline body surface area, from baseline to 12 months of treatment with finerenone compared to placebo.
Right Ventricular Ejection Fraction (RVEF) | 12 months
  Change in RVEF, measured by cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Right Ventricular End-Diastolic Volume indexed to baseline body surface area (RVEDVi) | 12 months
  Change in RVEDVi, measured by cMRI and indexed to baseline body surface area, from baseline to 12 months of treatment with finerenone compared to placebo.
Right Ventricular End-Systolic Volume indexed to baseline body surface area (RVESVi) | 12 months
  Change in RVESVi, measured by cMRI and indexed to baseline body surface area, from baseline to 12 months of treatment with finerenone compared to placebo.
Left Atrial Volume indexed to baseline body surface area (LAVi) | 12 months
  Change in LAVi, measured by cMRI and indexed to baseline body surface area, from baseline to 12 months of treatment with finerenone compared to placebo.

OTHER OUTCOMES:
Focal and Diffuse Fibrosis | 12 months
  Effect on focal fibrosis (assessed by late gadolinium enhancement and diffuse fibrosis (assessed by extracellular volume using T1 mapping) measured by cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - left ventricular global longitudinal strain | 12 months
  Effect on left ventricular global longitudinal strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - global circumferential strain | 12 months
  Effect on global circumferential strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - global radial strain | 12 months
  Effect on global radial strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - diastolic strain rate | 12 months
  Effect on diastolic strain rate, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - right ventricular free wall strain | 12 months
  Effect on right ventricular free wall strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - left atrial strain | 12 months
  Effect on left atrial strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
Myocardial Strain Parameters - right atrial strain | 12 months
  Effect on right atrial strain, assessed by speckle tracking echocardiography and/or feature-tracking cMRI, from baseline to 12 months of treatment with finerenone compared to placebo.
N-terminal pro-B-type natriuretic peptide (NT-proBNP) Levels | 12 months
  Change in NT-proBNP concentration from baseline to 12 months of treatment with finerenone compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — North York Diagnostic and Cardiac Centre
Locations (3):
- Canada (3):
  - Cambride Cardiac Care Centre, Cambridge, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Diagnostic Assessment Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Zhou R, Lu C, Chen Q, Xu T, Li D. Effects of the Angiotensin-Receptor Neprilysin Inhibitor on Cardiac Reverse Remodeling: Meta-Analysis. J Am Heart Assoc. 2019 Jul 2;8(13):e012272. doi: 10.1161/JAHA.119.012272. Epub 2019 Jun 26. PMID 31240976
- [Background] Santos-Gallego CG, Vargas-Delgado AP, Requena-Ibanez JA, Garcia-Ropero A, Mancini D, Pinney S, Macaluso F, Sartori S, Roque M, Sabatel-Perez F, Rodriguez-Cordero A, Zafar MU, Fergus I, Atallah-Lajam F, Contreras JP, Varley C, Moreno PR, Abascal VM, Lala A, Tamler R, Sanz J, Fuster V, Badimon JJ; EMPA-TROPISM (ATRU-4) Investigators. Randomized Trial of Empagliflozin in Nondiabetic Patients With Heart Failure and Reduced Ejection Fraction. J Am Coll Cardiol. 2021 Jan 26;77(3):243-255. doi: 10.1016/j.jacc.2020.11.008. Epub 2020 Nov 13. PMID 33197559
- [Background] Kasama S, Toyama T, Sumino H, Matsumoto N, Sato Y, Kumakura H, Takayama Y, Ichikawa S, Suzuki T, Kurabayashi M. Additive effects of spironolactone and candesartan on cardiac sympathetic nerve activity and left ventricular remodeling in patients with congestive heart failure. J Nucl Med. 2007 Dec;48(12):1993-2000. doi: 10.2967/jnumed.107.045427. Epub 2007 Nov 15. PMID 18006623
- [Background] Dorr K, Kammerlander A, Lauriero F, Lorenz M, Marculescu R, Beitzke D. Effect of etelcalcetide versus alfacalcidol on left ventricular function and feature-tracking cardiac magnetic resonance imaging in hemodialysis-a post-hoc analysis of a randomized, controlled trial. J Cardiovasc Magn Reson. 2023 Nov 6;25(1):62. doi: 10.1186/s12968-023-00975-4. PMID 37932788
- [Background] Everett RJ, Tastet L, Clavel MA, Chin CWL, Capoulade R, Vassiliou VS, Kwiecinski J, Gomez M, van Beek EJR, White AC, Prasad SK, Larose E, Tuck C, Semple S, Newby DE, Pibarot P, Dweck MR. Progression of Hypertrophy and Myocardial Fibrosis in Aortic Stenosis: A Multicenter Cardiac Magnetic Resonance Study. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007451. doi: 10.1161/CIRCIMAGING.117.007451. PMID 29914867
- [Background] Biederman RW, Magovern JA, Grant SB, Williams RB, Yamrozik JA, Vido DA, Rathi VK, Rayarao G, Caruppannan K, Doyle M. LV reverse remodeling imparted by aortic valve replacement for severe aortic stenosis; is it durable? A cardiovascular MRI study sponsored by the American Heart Association. J Cardiothorac Surg. 2011 Apr 14;6:53. doi: 10.1186/1749-8090-6-53. PMID 21492429
- [Background] Cicoira M, Zanolla L, Rossi A, Golia G, Franceschini L, Brighetti G, Marino P, Zardini P. Long-term, dose-dependent effects of spironolactone on left ventricular function and exercise tolerance in patients with chronic heart failure. J Am Coll Cardiol. 2002 Jul 17;40(2):304-10. doi: 10.1016/s0735-1097(02)01965-4. PMID 12106936
- [Background] Kosmala W, Przewlocka-Kosmala M, Szczepanik-Osadnik H, Mysiak A, Marwick TH. Fibrosis and cardiac function in obesity: a randomised controlled trial of aldosterone blockade. Heart. 2013 Mar;99(5):320-6. doi: 10.1136/heartjnl-2012-303329. Epub 2013 Jan 23. PMID 23343682
- [Background] Chan AK, Sanderson JE, Wang T, Lam W, Yip G, Wang M, Lam YY, Zhang Y, Yeung L, Wu EB, Chan WW, Wong JT, So N, Yu CM. Aldosterone receptor antagonism induces reverse remodeling when added to angiotensin receptor blockade in chronic heart failure. J Am Coll Cardiol. 2007 Aug 14;50(7):591-6. doi: 10.1016/j.jacc.2007.03.062. Epub 2007 Jul 30. PMID 17692742
- [Background] Vizzardi E, D'Aloia A, Giubbini R, Bordonali T, Bugatti S, Pezzali N, Romeo A, Dei Cas A, Metra M, Dei Cas L. Effect of spironolactone on left ventricular ejection fraction and volumes in patients with class I or II heart failure. Am J Cardiol. 2010 Nov 1;106(9):1292-6. doi: 10.1016/j.amjcard.2010.06.052. Epub 2010 Sep 9. PMID 21029826
- [Background] Verma S, Mazer CD, Yan AT, Mason T, Garg V, Teoh H, Zuo F, Quan A, Farkouh ME, Fitchett DH, Goodman SG, Goldenberg RM, Al-Omran M, Gilbert RE, Bhatt DL, Leiter LA, Juni P, Zinman B, Connelly KA. Effect of Empagliflozin on Left Ventricular Mass in Patients With Type 2 Diabetes Mellitus and Coronary Artery Disease: The EMPA-HEART CardioLink-6 Randomized Clinical Trial. Circulation. 2019 Nov 19;140(21):1693-1702. doi: 10.1161/CIRCULATIONAHA.119.042375. Epub 2019 Aug 22. PMID 31434508
- [Background] Zhou D, Huang Y, Cai A, Yan M, Cheng Q, Feng X, Nie Z, Feng Y. Longitudinal Study of Left Ventricular Mass Index Trajectories and Risk of Mortality in Hypertension: A Cohort Study. J Am Heart Assoc. 2023 May 2;12(9):e028568. doi: 10.1161/JAHA.122.028568. Epub 2023 Apr 29. PMID 37119065
- [Background] Verma A, Meris A, Skali H, Ghali JK, Arnold JM, Bourgoun M, Velazquez EJ, McMurray JJ, Kober L, Pfeffer MA, Califf RM, Solomon SD. Prognostic implications of left ventricular mass and geometry following myocardial infarction: the VALIANT (VALsartan In Acute myocardial iNfarcTion) Echocardiographic Study. JACC Cardiovasc Imaging. 2008 Sep;1(5):582-91. doi: 10.1016/j.jcmg.2008.05.012. PMID 19356485
- [Background] Rosch S, Kresoja KP, Besler C, Fengler K, Schober AR, von Roeder M, Lucke C, Gutberlet M, Klingel K, Thiele H, Rommel KP, Lurz P. Characteristics of Heart Failure With Preserved Ejection Fraction Across the Range of Left Ventricular Ejection Fraction. Circulation. 2022 Aug 16;146(7):506-518. doi: 10.1161/CIRCULATIONAHA.122.059280. Epub 2022 Jul 8. PMID 35862208
- [Background] Playford D, Strange G, Joseph M, Perry R, Chan YK, Strom JB, Spetko N, Harris SA, Stewart S, Selvanayagam JB. Increasing Left Ventricular Mass and Death in Men and Women Investigated With Echocardiography. J Am Heart Assoc. 2025 Dec 16;14(24):e041927. doi: 10.1161/JAHA.125.041927. Epub 2025 Dec 11. PMID 41378460
- [Background] Maki KC, Wilcox ML, Dicklin MR, Kakkar R, Davidson MH. Left ventricular mass regression, all-cause and cardiovascular mortality in chronic kidney disease: a meta-analysis. BMC Nephrol. 2022 Jan 16;23(1):34. doi: 10.1186/s12882-022-02666-1. PMID 35034619
- [Background] Laukkanen JA, Khan H, Kurl S, Willeit P, Karppi J, Ronkainen K, Di Angelantonio E. Left ventricular mass and the risk of sudden cardiac death: a population-based study. J Am Heart Assoc. 2014 Nov 5;3(6):e001285. doi: 10.1161/JAHA.114.001285. PMID 25376188
- [Background] Kawel-Boehm N, Kronmal R, Eng J, Folsom A, Burke G, Carr JJ, Shea S, Lima JAC, Bluemke DA. Left Ventricular Mass at MRI and Long-term Risk of Cardiovascular Events: The Multi-Ethnic Study of Atherosclerosis (MESA). Radiology. 2019 Oct;293(1):107-114. doi: 10.1148/radiol.2019182871. Epub 2019 Aug 27. PMID 31453766
- [Background] Gehlken C, Screever EM, Suthahar N, van der Meer P, Westenbrink BD, Coster JE, Van Veldhuisen DJ, de Boer RA, Meijers WC. Left atrial volume and left ventricular mass indices in heart failure with preserved and reduced ejection fraction. ESC Heart Fail. 2021 Aug;8(4):2458-2466. doi: 10.1002/ehf2.13366. Epub 2021 Jun 4. PMID 34085774
- [Background] Devereux RB, Wachtell K, Gerdts E, Boman K, Nieminen MS, Papademetriou V, Rokkedal J, Harris K, Aurup P, Dahlof B. Prognostic significance of left ventricular mass change during treatment of hypertension. JAMA. 2004 Nov 17;292(19):2350-6. doi: 10.1001/jama.292.19.2350. PMID 15547162
- [Background] de Simone G, Gottdiener JS, Chinali M, Maurer MS. Left ventricular mass predicts heart failure not related to previous myocardial infarction: the Cardiovascular Health Study. Eur Heart J. 2008 Mar;29(6):741-7. doi: 10.1093/eurheartj/ehm605. Epub 2008 Jan 19. PMID 18204091
- [Background] Brown LAE, Wahab A, Ikongo E, Saunderson CED, Jex N, Thirunavukarasu S, Chowdhary A, Das A, Craven TP, Levelt E, Dall'Armellina E, Knott KD, Greenwood JP, Moon JC, Xue H, Kellman P, Plein S, Swoboda PP. Cardiovascular magnetic resonance phenotyping of heart failure with mildly reduced ejection fraction. Eur Heart J Cardiovasc Imaging. 2022 Dec 19;24(1):38-45. doi: 10.1093/ehjci/jeac204. PMID 36285884
- [Background] Anstey DE, Tanner RM, Booth JN 3rd, Bress AP, Diaz KM, Sims M, Ogedegbe G, Muntner P, Abdalla M. Inappropriate Left Ventricular Mass and Cardiovascular Disease Events and Mortality in Blacks: The Jackson Heart Study. J Am Heart Assoc. 2019 Aug 20;8(16):e011897. doi: 10.1161/JAHA.118.011897. Epub 2019 Aug 13. PMID 31407619
- [Background] Gaasch WH, Zile MR. Left ventricular structural remodeling in health and disease: with special emphasis on volume, mass, and geometry. J Am Coll Cardiol. 2011 Oct 18;58(17):1733-40. doi: 10.1016/j.jacc.2011.07.022. PMID 21996383
- [Background] Zhang Y, Zhang X, Wang Y, Hu X, Wang B, Yang J, Zhao X, Zhang L. Relationship between diffuse fibrosis assessed by CMR and depressed myocardial strain in different stages of heart failure. Eur J Radiol. 2023 Jul;164:110848. doi: 10.1016/j.ejrad.2023.110848. Epub 2023 Apr 26. PMID 37156180
- [Background] Schelbert EB, Fridman Y, Wong TC, Abu Daya H, Piehler KM, Kadakkal A, Miller CA, Ugander M, Maanja M, Kellman P, Shah DJ, Abebe KZ, Simon MA, Quarta G, Senni M, Butler J, Diez J, Redfield MM, Gheorghiade M. Temporal Relation Between Myocardial Fibrosis and Heart Failure With Preserved Ejection Fraction: Association With Baseline Disease Severity and Subsequent Outcome. JAMA Cardiol. 2017 Sep 1;2(9):995-1006. doi: 10.1001/jamacardio.2017.2511. PMID 28768311
- [Background] Garg P, Assadi H, Jones R, Chan WB, Metherall P, Thomas R, van der Geest R, Swift AJ, Al-Mohammad A. Left ventricular fibrosis and hypertrophy are associated with mortality in heart failure with preserved ejection fraction. Sci Rep. 2021 Jan 12;11(1):617. doi: 10.1038/s41598-020-79729-6. PMID 33436786
- [Background] von Knobelsdorff-Brenkenhoff F, Schulz-Menger J. Role of cardiovascular magnetic resonance in the guidelines of the European Society of Cardiology. J Cardiovasc Magn Reson. 2016 Jan 22;18:6. doi: 10.1186/s12968-016-0225-6. PMID 26800662
- [Background] Karamitsos TD, Arvanitaki A, Karvounis H, Neubauer S, Ferreira VM. Myocardial Tissue Characterization and Fibrosis by Imaging. JACC Cardiovasc Imaging. 2020 May;13(5):1221-1234. doi: 10.1016/j.jcmg.2019.06.030. Epub 2019 Sep 18. PMID 31542534
- [Background] Haaf P, Garg P, Messroghli DR, Broadbent DA, Greenwood JP, Plein S. Cardiac T1 Mapping and Extracellular Volume (ECV) in clinical practice: a comprehensive review. J Cardiovasc Magn Reson. 2016 Nov 30;18(1):89. doi: 10.1186/s12968-016-0308-4. PMID 27899132
- [Background] Gupta S, Ge Y, Singh A, Grani C, Kwong RY. Multimodality Imaging Assessment of Myocardial Fibrosis. JACC Cardiovasc Imaging. 2021 Dec;14(12):2457-2469. doi: 10.1016/j.jcmg.2021.01.027. Epub 2021 May 19. PMID 34023250
- [Background] Ambale-Venkatesh B, Lima JA. Cardiac MRI: a central prognostic tool in myocardial fibrosis. Nat Rev Cardiol. 2015 Jan;12(1):18-29. doi: 10.1038/nrcardio.2014.159. Epub 2014 Oct 28. PMID 25348690
- [Background] Ali ND, Behairy N, Kharabish A, Elmozy W, Hegab AY, Saraya S. Cardiac MRI T1 mapping and extracellular volume application in hypertrophic cardiomyopathy. Egypt J Radiol Nucl Med. 2021;52:58.
- [Background] Unlu S, Ozden O, Celik A. Imaging in Heart Failure with Preserved Ejection Fraction: A Multimodality Imaging Point of View. Card Fail Rev. 2023 Apr 4;9:e04. doi: 10.15420/cfr.2022.27. eCollection 2023. PMID 37387734
- [Background] Rajiah PS, Francois CJ, Leiner T. Cardiac MRI: State of the Art. Radiology. 2023 May;307(3):e223008. doi: 10.1148/radiol.223008. Epub 2023 Apr 11. PMID 37039684
- [Background] Liu C, Ferrari VA, Han Y. Cardiovascular Magnetic Resonance Imaging and Heart Failure. Curr Cardiol Rep. 2021 Mar 8;23(4):35. doi: 10.1007/s11886-021-01464-9. PMID 33686516
- [Background] Han Y, Chen Y, Ferrari VA. Contemporary Application of Cardiovascular Magnetic Resonance Imaging. Annu Rev Med. 2020 Jan 27;71:221-234. doi: 10.1146/annurev-med-041818-015923. PMID 31986088
- [Background] Assadi H, Jones R, Swift AJ, Al-Mohammad A, Garg P. Cardiac MRI for the prognostication of heart failure with preserved ejection fraction: A systematic review and meta-analysis. Magn Reson Imaging. 2021 Feb;76:116-122. doi: 10.1016/j.mri.2020.11.011. Epub 2020 Nov 19. PMID 33221422
- [Background] Smiseth OA, Morris DA, Cardim N, Cikes M, Delgado V, Donal E, Flachskampf FA, Galderisi M, Gerber BL, Gimelli A, Klein AL, Knuuti J, Lancellotti P, Mascherbauer J, Milicic D, Seferovic P, Solomon S, Edvardsen T, Popescu BA; Reviewers: This document was reviewed by members of the 2018-2020 EACVI Scientific Documents Committee. Multimodality imaging in patients with heart failure and preserved ejection fraction: an expert consensus document of the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2022 Jan 24;23(2):e34-e61. doi: 10.1093/ehjci/jeab154. PMID 34729586
- [Background] Delcayre C, Silvestre JS, Garnier A, Oubenaissa A, Cailmail S, Tatara E, Swynghedauw B, Robert V. Cardiac aldosterone production and ventricular remodeling. Kidney Int. 2000 Apr;57(4):1346-51. doi: 10.1046/j.1523-1755.2000.00973.x. PMID 10760065
- [Background] Okoshi MP, Yan X, Okoshi K, Nakayama M, Schuldt AJ, O'Connell TD, Simpson PC, Lorell BH. Aldosterone directly stimulates cardiac myocyte hypertrophy. J Card Fail. 2004 Dec;10(6):511-8. doi: 10.1016/j.cardfail.2004.03.002. PMID 15599842
- [Background] Brilla CG, Weber KT. Mineralocorticoid excess, dietary sodium, and myocardial fibrosis. J Lab Clin Med. 1992 Dec;120(6):893-901. PMID 1453111
- [Background] Tanabe A, Naruse M, Naruse K, Hase M, Yoshimoto T, Tanaka M, Seki T, Demura R, Demura H. Left ventricular hypertrophy is more prominent in patients with primary aldosteronism than in patients with other types of secondary hypertension. Hypertens Res. 1997 Jun;20(2):85-90. doi: 10.1291/hypres.20.85. PMID 9220271
- [Background] Rossi GP, Di Bello V, Ganzaroli C, Sacchetto A, Cesari M, Bertini A, Giorgi D, Scognamiglio R, Mariani M, Pessina AC. Excess aldosterone is associated with alterations of myocardial texture in primary aldosteronism. Hypertension. 2002 Jul;40(1):23-7. doi: 10.1161/01.hyp.0000023182.68420.eb. PMID 12105133
- [Background] Buffolo F, Tetti M, Mulatero P, Monticone S. Aldosterone as a Mediator of Cardiovascular Damage. Hypertension. 2022 Sep;79(9):1899-1911. doi: 10.1161/HYPERTENSIONAHA.122.17964. Epub 2022 Jun 29. PMID 35766038
- See also: American Heart Association Inc. Classes and Stages of Heart Failure. American Heart Association. — https://www.heart.org/en/health-topics/heart-failure/what-is-heart-failure/classes-of-heart-failure